CLINICAL TRIAL: NCT06924957
Title: Influence of Body Position on the Defecation Model Measured During High Resolution Anorectal Manometry in Children- a Control Study.
Brief Title: Influence of Body Position on the Defecation Model During Anorectal Manometry.
Acronym: HRAMposition
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Marcin Banasiuk, MD PhD, Medical University of Warsaw
Other Study IDs: Banasiuk2021B
Record Dates: First submitted 2024-11-12; First posted 2025-04-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Constipation; Children; Anorectal Disorder
Keywords: anorectal manometry; HRAM; constipasion; position
MeSH Terms: conditions — Constipation; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Constipation group: Children that meet Rome IV criteria to diagnose functional constipation.
  Interventions: Other: 3D HRAM
- Healthy volounteers: Children without IBD, without chronic diseases of GI tract nor history of anorectal surgery
  Interventions: Other: 3D HRAM

INTERVENTIONS:
Other: 3D HRAM — The test will be performed both in supine and sitting position successively, using 3D HR-ARM. Resting, squeeze pressures, and bear down manoeuvre variables will be obtained. Diagnosis of dyssynergic defecation requires < 20% relaxation of anal sphincter and/or intrarectal pressure>40 mmHg during bear down manoeuvre.
  Other Names: Three-dimensional high-resolution anorectal manometry

SUMMARY:
Anorectal 3D manometry (3D HRAM) is the most advanced version of manometric equipment that measures pressures along the anal canal in a very detailed manner. It provides complete data about pressure profile of anorectum and may indicate impaired defecation dynamics. Resent studies suggest that the position in which 3D HRAM is performed should be changed. So far, no scientific research has been performed in children that directly compares both positions. The reference values of registered pressures during 3D HRAM in people without complaints were not specified, which would allow for a more precise diagnosis of patients with an incorrect defecation model and precise selection of patients who could benefit from biofeedback therapy.

DETAILED DESCRIPTION:
Patients with the diagnosis of constipation will be enrolled in the study. Each patient will be investigated by anorectal manometry in both- sitted and lying position.

During anorectal manometry conventional manometric parameters will be recorded, such as resting pressure, squeeze pressure, bear down manoeuver, thresholds of sensation and threshold of recto anal inhibitory reflex. 3D picture of anal canal will be recorded.

ELIGIBILITY:
Inclusion criteria - the study group:

* age from 5 to 18 years old
* functional constipation diagnosed on the basis of Rome IV criteria
* parental or guardian written consent to the participation of the child in the study; in the case of a child ≥16 years old also the child's written consent

Inclusion criteria - the control group:

* age from 5 to 18 years old
* no lower gastrointestinal symptoms
* parental or guardian written consent to the participation of the child in the study; in the case of a child ≥16 years old also the child's written consent

Exclusion criteria - the study group and the control group:

* undergone surgeries due to congenital anomalies in the lower gastrointestinal tract
* inflammatory bowel diseases or inflammation of the large intestine with a different aetiology
* anal fissure, inflammation of the anal area or other conditions which, in the opinion of the researcher, could affect the functioning of the distal gastrointestinal tract

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample size was calculated to detect a 45% difference in the percentage of patients with a negative rectoanal gradient, assuming equal groups, alpha = 0.05, beta = 0.1, and a 30% drop out percentage. There should be 30 people in the constipation group and 30 healthy volunteers.
  Due to possible differences depending on age, it was decided to conduct the study in two separate age groups (I. younger, i.e. 5-10 years old and II. older, 11-18 years old). The total number of patients in the study will therefore be 120 people.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DD frequency | 1 day
  The difference in the number of patients with DD (defined as <20% relaxation of anal sphincter and/or intrarectal pressure >40 mmHg during bear down manoeuvre) in sitting and lying position.

SECONDARY OUTCOMES:
Values of pressures obtained during anorectal manometry | 1 day
  Values of manometric parameters obtained in the lying and sitting position: mean resting pressure of the anal sphincter (mmHg), maximum squeeze pressure (mmHg), residual anal pressure (mmHg).
Values of mean anal canal length | 1 day
  The mean anal canal length will be assessed in sitting and lying position in the two groups.
Percentage of anal relaxation rate | 1 day
  the assessment of parameters of defecation dynamics during HR-ARM: rectoanal pressure gradient. All secondary end points will be assessed in sitting and lying position in the two groups.
  the assessment of parameters of defecation dynamics during HR-ARM: percentage of anal relaxation rate, rectoanal pressure gradient. All secondary

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Skowrońska, MD, Principal Investigator — Department of Pediatric Gastroenterology Medical University of Warsaw
Locations (1):
- The Department of Paediatric Gastroenterology and Nutrition, Warsaw Medical University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SS, Kavlock R, Rao S. Influence of body position and stool characteristics on defecation in humans. Am J Gastroenterol. 2006 Dec;101(12):2790-6. doi: 10.1111/j.1572-0241.2006.00827.x. Epub 2006 Oct 6. PMID 17026568
- [Background] Su H, Peng LH, Sun G, Yang YS, Wu J, Jiang GJ, Ge H. Effect of different body position on anorectal manometry for chronic constipation patients. Eur Rev Med Pharmacol Sci. 2019 Oct;23(19):8493-8500. doi: 10.26355/eurrev_201910_19162. PMID 31646580
- [Background] Wu GJ, Xu F, Lin L, Pasricha PJ, Chen JDZ. Anorectal manometry: Should it be performed in a seated position? Neurogastroenterol Motil. 2017 May;29(5). doi: 10.1111/nmo.12997. Epub 2016 Dec 1. PMID 27910245
- [Background] Coss-Adame E, Rao SS, Valestin J, Ali-Azamar A, Remes-Troche JM. Accuracy and Reproducibility of High-definition Anorectal Manometry and Pressure Topography Analyses in Healthy Subjects. Clin Gastroenterol Hepatol. 2015 Jun;13(6):1143-50.e1. doi: 10.1016/j.cgh.2014.12.034. Epub 2015 Jan 20. PMID 25616028
- [Background] Grossi U, Carrington EV, Bharucha AE, Horrocks EJ, Scott SM, Knowles CH. Diagnostic accuracy study of anorectal manometry for diagnosis of dyssynergic defecation. Gut. 2016 Mar;65(3):447-55. doi: 10.1136/gutjnl-2014-308835. Epub 2015 Mar 12. PMID 25765461
- [Derived] Skowronska B, Banaszkiewicz A, Banasiuk M. Influence of body position on defecation mechanics measured during high-resolution anorectal manometry in paediatric population: a protocol for case-control study. BMJ Open. 2025 Dec 31;15(12):e112928. doi: 10.1136/bmjopen-2025-112928. PMID 41475818

DOCUMENTS (2):
  • Study Protocol (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06924957/Prot_000.pdf
  • Informed Consent Form (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT06924957/ICF_001.pdf